CLINICAL TRIAL: NCT04224467
Title: Real-Time Identification of Lesions and Nerves by Using Indocyanine Green Fluorescent Imaging in Gynecological Surgery
Brief Title: The Application of Real-Time Near-infrared Imaging in Gynecological Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chen Chunlin (Other)
Collaborators: Chinese Academy of Sciences (Other Government)
Responsible Party: Sponsor-Investigator, Chen Chunlin, Department of Obstetrics and Gynecology, Southern Medical University, China
Organization: Southern Medical University, China (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NFEC-2019-242
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Cervical Cancer; Ovarian Tumor; Endometrial Carcinoma; Uterine Myomatosis; Adenomyosis; Ovarian Cyst Benign; Ovarian Cyst Malignant; Endometriosis; Uterine Sarcoma
MeSH Terms: conditions — Uterine Cervical Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms; Adenomyosis; Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Indocyanine Green Fluorescent Imaging (Experimental): Patients will be intravenously injected ICG (Yichuang Pharmaceutical Limited Liability Company, Dandong, China) at a dose of 2-5 mg per kg of body weight before surgery or 0.25-0.5 mg per kg of body weight during surgery. Then, a NIR imaging systems included the NIR (800-900 nm) and white-light (400-650nm) dual-channel will be used to detect In situ lesions, metastatic lesions, lymph nodes, obturator nerve, pelvic autonomic nerve, etc during surgery according to disease and clinical needs.
  Interventions: Other: Intravenous ICG and Real-Time Near-infrared Imaging

INTERVENTIONS:
Other: Intravenous ICG and Real-Time Near-infrared Imaging — Patients will be intravenously injected ICG (Yichuang Pharmaceutical Limited Liability Company, Dandong, China) at a dose of 2-5 mg per kg of body weight before surgery or 0.25-0.5 mg per kg of body weight during surgery. Then real-time near-infrared imaging will be conducted during surgery.

SUMMARY:
Removing in situ and metastasis lesions completely during gynecological surgery is central to reduce the recurrence and death, and the identification of lesions in traditional gynecological surgery often depends on the experience of surgeons. The identification of nerves is often needed in gynecological surgery, such as the obturator nerves in pelvic lymphadenectomy, and the pelvic autonomic nerves in nerve-sparing radical hysterectomy for cervical cancer. Nerve identification also relies heavily on the experience of surgeons. This project aims to realize the identification of lesions and nerves under the navigation of indocyanine green fluorescent imaging, and evaluate the accuracy of fluorescent imaging of lesions and the effectiveness of nerves identification by near-infrared imaging. This project may reduce the recurrence or death caused by residual lesions and postoperative dysfunction caused by nerves injury, thus, improve the survival rate and quality of life for patients with gynecological diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients with FIGO (2018) stage IA1(LVSI)-IIA2 cervical cancer，endometrial cancer，ovarian tumor, endometriosis, adenomyosis, uterine myomatosis, ovarian cyst ,or uterine sarcoma
* Patients who consent to receive indocyanine green near-infrared fluorescence-guided gynecological surgery

Exclusion Criteria:

* Less than 6 months expectancy life;
* Patients with iodine allergy.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
The value and feasibility of real-time near-infrared imaging in the identification of lesions | 4 years
  Evaluation of the effectiveness of real-time near-infrared imaging in detecting the margin of in situ lesions, whether there is metastasis lesions and whether the metastasis lesions has been completely removed , lymph node metastasis or not during gynecological surgery. The criteria of evaluation is postoperative pathological results and fluorescence intensity of specimen sections measured by laser scanning confocal microscope.
The value and feasibility of real-time near-infrared imaging in the identification of nerves | 4 years
  Evaluation of the effectiveness of real-time near-infrared imaging in detecting nerves associated with gynecological surgery, including the pelvic autonomic nerves composed of the abdominal aortic plexus, the superior hypogastric plexus, the hypogastric nerves, the pelvic splanchnic nerves, the inferior hypogastric plexus and its branches, obturator nerves, genitofemoral nerve, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Southern Medical Universtity, China, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Seracchioli R, Raimondo D, Arena A, Zanello M, Mabrouk M. Clinical use of endovenous indocyanine green during rectosigmoid segmental resection for endometriosis. Fertil Steril. 2018 Jun;109(6):1135. doi: 10.1016/j.fertnstert.2018.02.122. PMID 29935649
- [Result] Gossedge G, Vallance A, Jayne D. Diverse applications for near infra-red intraoperative imaging. Colorectal Dis. 2015 Oct;17 Suppl 3:7-11. doi: 10.1111/codi.13023. PMID 26394736
- [Result] Cosentino F, Vizzielli G, Turco LC, Fagotti A, Cianci S, Vargiu V, Zannoni GF, Ferrandina G, Scambia G. Near-Infrared Imaging with Indocyanine Green for Detection of Endometriosis Lesions (Gre-Endo Trial): A Pilot Study. J Minim Invasive Gynecol. 2018 Nov-Dec;25(7):1249-1254. doi: 10.1016/j.jmig.2018.02.023. Epub 2018 Mar 15. PMID 29551477
- [Result] Malzoni M, Iuzzolino D, Rasile M, Coppola M, Casarella L, Di Giovanni A, Falcone F. Surgical Principles of Segmental Rectosigmoid Resection and Reanastomosis for Deep Infiltrating Endometriosis. J Minim Invasive Gynecol. 2020 Feb;27(2):258. doi: 10.1016/j.jmig.2019.06.018. Epub 2019 Jul 17. PMID 31325591
- [Result] He K, Zhou J, Yang F, Chi C, Li H, Mao Y, Hui B, Wang K, Tian J, Wang J. Near-infrared Intraoperative Imaging of Thoracic Sympathetic Nerves: From Preclinical Study to Clinical Trial. Theranostics. 2018 Jan 1;8(2):304-313. doi: 10.7150/thno.22369. eCollection 2018. PMID 29290809
- [Result] Chen SC, Wang MC, Wang WH, Lee CC, Yang TF, Lin CF, Wang JT, Liao CH, Chang CC, Chen MH, Shih YH, Hsu SP. Fluorescence-assisted visualization of facial nerve during mastoidectomy: A novel technique for preventing iatrogenic facial paralysis. Auris Nasus Larynx. 2015 Apr;42(2):113-8. doi: 10.1016/j.anl.2014.08.008. Epub 2014 Sep 6. PMID 25199746
- [Result] Mao Y, Chi C, Yang F, Zhou J, He K, Li H, Chen X, Ye J, Wang J, Tian J. The identification of sub-centimetre nodules by near-infrared fluorescence thoracoscopic systems in pulmonary resection surgeries. Eur J Cardiothorac Surg. 2017 Dec 1;52(6):1190-1196. doi: 10.1093/ejcts/ezx207. PMID 28950327
- [Derived] Li P, Liu J, He K, Gong S, Chi C, Liu P, Su G, Li W, Duan H, Liu P, Tian J, Chen C. Tumor lesion detection in patients with cervical cancer by indocyanine green near-infrared imaging. Eur J Nucl Med Mol Imaging. 2023 Mar;50(4):1252-1261. doi: 10.1007/s00259-022-06030-1. Epub 2022 Dec 1. PMID 36450938
- [Derived] He K, Li P, Zhang Z, Liu J, Liu P, Gong S, Chi C, Liu P, Chen C, Tian J. Intraoperative near-infrared fluorescence imaging can identify pelvic nerves in patients with cervical cancer in real time during radical hysterectomy. Eur J Nucl Med Mol Imaging. 2022 Jul;49(8):2929-2937. doi: 10.1007/s00259-022-05686-z. Epub 2022 Mar 1. PMID 35230489